CLINICAL TRIAL: NCT06789471
Title: The Effects of Psyllium Seed on Body Weight and Metabolic Syndrome Indicators in Patients
Brief Title: The Effects of Psyllium Seed on Body Weight and Metabolic Syndrome Indicators in Patients with Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ru-Shin Zhang (Other)
Responsible Party: Sponsor-Investigator, Ru-Shin Zhang, Taichung Hospital Nurse Practitioner, Hung Kaung University
Organization: Hung Kaung University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 112033
Record Dates: First submitted 2024-12-23; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-11

CONDITIONS: Overweight and Obesity; Metabolic Cardiovascular Syndrome; Schizophrenia, Disorganized
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome; Schizophrenia, Disorganized | interventions — Psyllium

STUDY DESIGN:
Intervention Model Description: . This study will be matched based on gender, age (within 10 years), and the same hospital.The participants will be divided into two groups using a single-masked randomized allocation method. The experimental group (psyllium husk group) will consume 10 grams of psyllium husk daily, divided into two doses, and taken approximately one hour before meals. The control group will receive standard treatment, and the intervention will last for 12 weeks. Inclusion criteria are: 1. Diagnosis of schizophrenia based on DSM-V criteria; 2. Age between 20 and 65 years old; 3. Body mass index (BMI) of 24 kg/m² or higher or those who meet more than three indicators of metabolic syndrome. Exclusion criteria are medications for lowering blood glucose, blood pressure, or lipid levels, significant comorbidities such as cardiovascular diseases or cancer, history of neurogenic bowel obstruction or post-weight loss surgery, and patients with prominent psychiatric symptoms who cannot cooperate.
Who Masked: Care Provider
Masking Description: single-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psyllium group (Experimental): The experimental group (psyllium husk group) will consume 10 grams of psyllium husk daily, divided into two doses, and taken approximately one hour before meals for 12 weeks.
  Interventions: Dietary Supplement: psyllium husk
- Control group (No Intervention): The control group will receive standard treatment, not use psyllium and the intervention will last for 12 weeks.

INTERVENTIONS:
Dietary Supplement: psyllium husk — Psyllium husk, derived from the seeds' husks of the Plantago ovata plant, is a plant-based fiber supplement.
  Arms: Psyllium group

SUMMARY:
The research employs a quasi-experimental design, aiming to enroll 24 hospitalized patients with schizophrenia from 2hospitals in the central region, guided by G Power calculations. Participants will be carefully matched based on gender, age (within 5 years), and the same hospital. They will be divided into two groups using a single-masked randomized allocation method. The experimental group (psyllium husk group) will consume 10 grams of psyllium husk daily, split into two doses, taken about an hour before meals. The control group will receive standard treatment. The intervention will last for 12 weeks.

Inclusion criteria involve a schizophrenia diagnosis as per DSM-V criteria, age between 20 and 65 years, and a body mass index (BMI) of 24 kg/m² or higher, or meeting more than three indicators of metabolic syndrome. Exclusion criteria include medications for glucose, blood pressure, or lipid levels reduction, significant comorbidities like cardiovascular diseases or cancer, a history of neurogenic bowel obstruction or post-weight loss surgery, and patients with severe psychiatric symptoms impeding cooperation.

Each patient will undergo measurements for weight, waist circumference, body mass index, and blood biochemical analysis, encompassing fasting blood glucose (FBG), total cholesterol (TC), triglycerides (TG), high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), and glycated hemoglobin (HbA1c) before the intervention and after 12 weeks.

DETAILED DESCRIPTION:
The study adopts a quasi-experimental research design and plans to include 24 hospitalized patients with schizophrenia from 2 hospitals in the central region, based on G Power calculations. This study will be matched based on gender, age (within 10 years), and the same hospital.The participants will be divided into two groups using a single-masked randomized allocation method. The experimental group (psyllium husk group) will consume 10 grams of psyllium husk daily, divided into two doses, and taken approximately one hour before meals. The control group will receive standard treatment, and the intervention will last for 12 weeks. Inclusion criteria are: 1. Diagnosis of schizophrenia based on DSM-V criteria; 2. Age between 20 and 65 years old; 3. Body mass index (BMI) of 24 kg/m² or higher or those who meet more than three indicators of metabolic syndrome. Exclusion criteria are medications for lowering blood glucose, blood pressure, or lipid levels, significant comorbidities such as cardiovascular diseases or cancer, history of neurogenic bowel obstruction or post-weight loss surgery, and patients with prominent psychiatric symptoms who cannot cooperate. Each patient will undergo measurements of weight, waist circumference, body mass index, and blood biochemical analysis data, including fasting blood glucose (FBG), total cholesterol (TC), triglycerides (TG), high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), and glycated hemoglobin (HbA1c) before the intervention and after 12 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of schizophrenia based on DSM-V criteria;
2. Age between 20 and 65 years old
3. Body mass index (BMI) of 24 kg/m² or higher or those who meet more than three indicators of metabolic syndrome
4. Individuals with glycated hemoglobin (HbA1c) levels ranging from 5.7% to 6.4%.

Exclusion Criteria:

1. Exclude those who use blood sugar-lowering, blood pressure-lowering, and blood-lipid-lowering drugs.
2. Patients with major internal and external diseases such as cardiovascular disease, cancer, patients who have experienced neuropathic intestinal obstruction, patients after bariatric surgery, or those who have experienced choking.
3. Those with obvious mental symptoms who are unable to cooperate.
4. History of grain allergy, asthma, etc.
5. Persons subject to a declaration of auxiliary guardianship.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Men and women aged between 20 and 65 years old
Enrollment: 24 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Body Weight in Kilograms | At baseline (week 0) and at weeks 6 and 12 of the study.
  Measure body weight in the morning after waking up, with participants wearing light clothing and no shoes.
Waist Circumference in cm | At baseline (week 0) and at weeks 6 and 12 of the study.
  Waist circumference will be measured to evaluate the impact of psyllium husk intervention on abdominal fat distribution in patients with schizophrenia. Measurements will be conducted using a flexible, non-stretchable measuring tape, positioned horizontally around the abdomen at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest. Participants will stand upright, with feet close together, arms at their sides, and abdomen relaxed during the measurement. The values will be recorded in centimeters (cm). The experimental group will consume 10 grams of psyllium husk daily, while the control group will receive standard treatment. Changes in waist circumference will be analyzed within and between groups."
Body Mass Index (BMI) in (kg/m²) | At baseline (week 0) and at weeks 6 and 12 of the study.
  Body mass index (BMI) will be calculated to evaluate the impact of psyllium husk intervention on overall body composition in patients with schizophrenia. BMI is expressed in kilograms per square meter (kg/m²) and will be calculated using the formula: weight (kg) divided by height squared (m²). Weight will be measured with a calibrated digital scale, ensuring participants wear light clothing and no shoes. Height will be measured using a wall-mounted stadiometer, with participants standing barefoot, heels together, arms at their sides, and head positioned in the Frankfurt horizontal plane. These measurements will be used to calculate BMI, which will be recorded and analyzed for changes within and between groups.

SECONDARY OUTCOMES:
Metabolic syndrome indicators ex (Fasting Glucose (mg/dL) Total Cholesterol (mg/dL) Triglycerides (mg/dL) High-Density Lipoprotein Cholesterol (HDL-C, mg/dL) Low-Density Lipoprotein Cholesterol (LDL-C, mg/dL) Glycated Hemoglobin (HbA1c, %) | During weeks 0 and 12of the study
  Each time, 5 c.c. of blood is drawn from the arm vein for the following tests and their respective units:
  Fasting Glucose (mg/dL) Total Cholesterol (mg/dL) Triglycerides (mg/dL) High-Density Lipoprotein Cholesterol (HDL-C, mg/dL) Low-Density Lipoprotein Cholesterol (LDL-C, mg/dL) Glycated Hemoglobin (HbA1c, %) Blood collection requires at least 8 hours of fasting and is performed by professional medical technologists or nursing staff to ensure accurate results.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Ling Lin, Study Director — HungKaungUniversity
Locations (1):
- Taichung Hospital, Taichung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No